CLINICAL TRIAL: NCT06144567
Title: Ultrasound-based Response of Enthesitis to Upadacitinib in Psoriatic Arthritis
Brief Title: Response to Upadacitinib of Enthesitis Evaluated by Ultrasound in Patients With Psoriatic Arthritis
Status: Not yet recruiting | Type: Observational
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Collaborators: Hospital Universitario de Móstoles (Other)
Responsible Party: Sponsor
Other Study IDs: A24- 391
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Psoriatic Arthritis
Keywords: Ultrasound; Entheses; Psoriatic arthritis; Upadacitinib
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — upadacitinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Adult patients with PsA according to CASPAR classification criteria: Adult patients (aged ≥ 18 years old and ≤ 65 years old) with PsA according to CASPAR classification criteria, who have been prescribed upadacitinib over the course of routine practice, in accordance with the applicable approved label and local regulatory and reimbursement policies ("In patients with psoriatic arthritis, upadacitinib would be a therapeutic alternative after failure, inadequate response or intolerance to csDMARDs and anti-TNF") and have at least one ultrasound-determined peripheral enthesitis.
  Interventions: Drug: Upadacitinib

INTERVENTIONS:
Drug: Upadacitinib — As this is an observational study, AbbVie is not involved in the product supply since the drug is being used according to the approved marketing label and is to be prescribed by the physician under usual and customary practice of physician prescription.
  Other Names: Rinvoq

SUMMARY:
Primary objective To evaluate the peripheral enthesitis response to upadacitinib treatment by BMUS and DMUS, in PsA patients at week 24.

Secondary objective:

1. To evaluate the peripheral enthesitis response to upadacitinib treatment by BMUS and DMUS, in PsA patients at week 12.
2. To evaluate the clinical response of enthesitis to upadacitinib by LEI, at week 12 and week 24.
3. To evaluate the clinical response of disease activity by DAPSA, at week 12 and week 24.

Study Design: single-arm, observational longitudinal, prospective study

Population: The study population will consist of adult patients (aged ≥ 18 years old and ≤ 65 years old) with PsA according to CASPAR classification criteria, who have been prescribed upadacitinib over the course of routine practice, in accordance with the applicable approved label and local regulatory and reimbursement policies ("In patients with psoriatic arthritis, upadacitinib would be a therapeutic alternative after failure, inadequate response or intolerance to csDMARDs and anti-TNF") and have at least one ultrasound-determined peripheral enthesitis.

DETAILED DESCRIPTION:
Rationale and Background:

Psoriatic arthritis (PsA) is a complex and heterogeneous skin-musculoskeletal disease with a broad clinical phenotype spectrum of mostly peripheral (i.e., arthritis, enthesitis, dactylitis) but also axial (i.e., spondylitis) manifestations. Among PsA domains, enthesitis in addition to being a hallmark of the disease, has shown to be associated with higher disease activity, disability, and incapacity to work, ultimately leading to poor quality of life. In clinical practice and clinical trials in PsA, enthesitis has traditionally been measured by physical examination or by clinical indices developed for spondyloarthritis (SpA), however, clinical examination of entheses depends on eliciting tenderness on direct palpation of the insertional site and may be not only nonspecific and insensitive, but also does not inform of the grade of inflammation or the presence of underlying structural changes. Ultrasound has clearly demonstrated higher sensitivity than clinical assessment for detecting enthesitis in PsA patients. Since 2008, under the umbrella of the Outcome Measures in Rheumatology (OMERACT) Ultrasound Group, a subtask force for enthesitis was created to produce standardized, agreed definitions of ultrasound-detected enthesitis components and a reliable scoring system for enthesitis.

Following a stepwise consensus-based methodology, the group agreed on the definitions of the elementary components of enthesitis and then decided which of them should be included in the final definition of an ultrasound-detected enthesitis for SpA/ PsA. Since 2014, through a number of consecutive live scanning exercises on patients with SpA and PsA, the intraobserver and interobserver reliability of the ultrasound elementary lesions and the scoring system of enthesitis was successfully tested. Furthermore, the responsiveness of ultrasound-determined enthesitis has been demonstrated in multicentre studies on patients with SpA/PsA treated with TNF inhibitors.

There are no studies on ultrasound-assessed enthesitis response to upadacitinib. In patients who have an inadequate response (IR) to conventional synthetic (cs) DMARDs in SELECT-PsA 1 clinical trial, both doses of upadacitinib demonstrated statistical differences versus placebo in clinical resolution of enthesitis according to LEI. In bDMARD-IR patients (SELECT-PsA 2), as an exploratory endpoint, a greater proportion of patients reached clinical resolution of enthesitis by LEI and SPARCC, on either dose of upadacitinib versus placebo. The results of the current ultrasound-based study will further characterize the effectiveness of upadacitinib in the enthesitis domain.

Primary objective To evaluate the peripheral enthesitis response to upadacitinib treatment by BMUS and DMUS, in PsA patients at week 24.

Secondary objective:

1. To evaluate the peripheral enthesitis response to upadacitinib treatment by BMUS and DMUS, in PsA patients at week 12.
2. To evaluate the clinical response of enthesitis to upadacitinib by LEI, at week 12 and week 24.
3. To evaluate the clinical response of disease activity by DAPSA, at week 12 and week 24.

Study Design: single-arm, observational longitudinal, prospective study

Population: The study population will consist of adult patients (aged ≥ 18 years old and ≤ 65 years old) with PsA according to CASPAR classification criteria, who have been prescribed upadacitinib over the course of routine practice, in accordance with the applicable approved label and local regulatory and reimbursement policies ("In patients with psoriatic arthritis, upadacitinib would be a therapeutic alternative after failure, inadequate response or intolerance to csDMARDs and anti-TNF") and have at least one ultrasound-determined peripheral enthesitis.

Variables:

Primary endpoint Changes from baseline in B-mode and Doppler-mode enthesitis measured by the OMERACT enthesitis scoring system at 24 weeks of follow-up.

Secondary endpoint Changes in B-mode and Doppler-mode enthesitis measured by the OMERACT enthesitis scoring system at 12 weeks.

Change in DAPSA score between baseline to week 12 and baseline to week 24. Change in LEI score between baseline to week 12 and baseline to week 24.

Descriptive variables (Baseline, 12 weeks, 24 weeks) Treatment for PsA Joint tenderness in 68 joints Joint swelling in 66 joints Patient's assessment of pain (NRS 0-10) Patient's Global Assessment of Disease Activity (PtGA) Psoriatic Arthritis Impact of Disease (PsAID12) SPARCC enthesitis index Presence of dactylitis in hands or feet C-reactive protein (CRP) Health Assessment Questionnaire-Disability Index (HAQ-DI)

Data Sources: Patient medical records, clinical and ultrasound assessments.

Study Size: 19 patients.

Data Analysis:

Categorical variables will be summarized with frequency and percentage. Continuous variables will be summarized with descriptive statistics (mean and standard deviation, median, minimum, and maximum); if these variables show a skewed distribution of values, median and interquartile range will also be reported.

Changes from baseline variation in the OMERACT enthesitis scoring, DAPSA, SPARCC and LEI score will be analysed by means of the Wilcoxon signed rank test for paired samples.

Correlations between clinical and BMUS/PDUS quantitative variables will be analysed using Spearman's correlation test. If association is demonstrated, it will be considered poor correlation if r < 0.2, fair correlation if r≥0.2 and r < 0.4, moderate correlation if r ≥0.4 and r < 0.7 and strong correlation if r ≥0.7.

Nominal p-value will be provided for associations.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female, at least ≥ 18 years old and ≤ 65 years old at Screening.
* Clinical diagnosis of PsA with symptom onset at least 6 months prior to the Screening visit and fulfillment of the Classification Criteria for PsA (CASPAR) (19).
* Physician decision on patient treatment with upadacitinib must have been reached prior to and independently of recruitment in the study.
* Upadacitinib prescribed in accordance with the applicable approved label and local regulatory and reimbursement policies.
* Inadequate response or intolerance to at least one bDMARD, one of them must be an anti-TNF according to the Spanish regulatory and reimbursement policies ("informe de posicionamiento terapéutico").
* Patients should have at least one ultrasound-determined peripheral enthesitis site according to OMERACT definition for ultrasound enthesitis.
* Subjects must voluntarily sign and date an informed consent.

Exclusion Criteria:

* Patients who cannot be treated with upadacitinib according to the approved label (e.g., contraindications).
* Consideration by the investigator, for any reason, that the subject is an unsuitable candidate to receive upadacitinib.
* Unwillingness or inability to comply with the study requirements.
* Prior exposure to any Janus kinase (JAK) inhibitor.
* Patients taking ≥ 10 mg of prednisone or equivalent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients (aged ≥ 18 years old and ≤ 65 years old) with PsA according to CASPAR classification criteria, who have been prescribed upadacitinib over the course of routine practice, in accordance with the applicable approved label and local regulatory and reimbursement policies ("In patients with psoriatic arthritis, upadacitinib would be a therapeutic alternative after failure, inadequate response or intolerance to csDMARDs and anti-TNF") and have at least one ultrasound-determined peripheral enthesitis site. The study plans to enroll 19 patients.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Changes in B-mode and Doppler-mode ultrasound enthesitis | Baseline to week 24
  Changes from baseline in B-mode and Doppler-mode enthesitis measured by the Outcome Meaures in Rheumatology (OMERACT) enthesitis scoring system (0, no to 3, severe, at each evaluated enthesis) at 24 weeks of follow-up.

SECONDARY OUTCOMES:
Changes in B-mode and Doppler-mode ultrasound enthesitis | Baseline to week12
  Changes in B-mode and Doppler-mode enthesitis measured by the OMERACT enthesitis scoring system at 12 weeks.
Change in Disease Activity in Psoriatic Arthritis (DAPSA) score | Baseline to week 12 ans 24
  Change in DAPSA score between baseline to week 12 and baseline to week 24.
Change in Leeds Enthesitis Index (LEI) score (0-6) | Baeline to week 12 ans 24
  Change in LEI score between baseline to week 12 and baseline to week 24.

CONTACTS AND LOCATIONS:
Overall Officials: Esperanza Naredo, Principal Investigator — Hospital Universitario Fundación Jiménez Díaz
Locations (1):
- Instituto de Investigación Sanitaria Fundación Jiménez Díaz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No